CLINICAL TRIAL: NCT00956735
Title: Effects of Pistachios on Cardiovascular Responses to Stress in Type 2 Diabetes: A Novel Intervention for a High Risk Population
Brief Title: Effects of Pistachios on Cardiovascular Responses to Stress in Type 2 Diabetes
Acronym: Pistachio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: American Pistachio Growers (Other)
Responsible Party: Principal Investigator, Sheila G West, Associate Professor, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 29970
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Cardiovascular Disease; Type 2 Diabetes
Keywords: Cardiovascular Disease; Type II Diabetes; Nutrition; Pistachios; Cardiovascular disease risk factors in adults with Type II diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pistachio Diet (Experimental): Incorporates 3.0 oz (2 servings) of pistachios into a daily diet
  Interventions: Other: Pistachio
- Non-Pistachio (No Intervention): Does not incorporate pistachios into a daily diet

INTERVENTIONS:
Other: Pistachio — 3.0 oz (2 servings) of roasted and salted or unsalted pistachios
  Arms: Pistachio Diet

SUMMARY:
This study is investigating the effects of three different diets, including a diet with pistachios, on cardiovascular disease risk markers in people with type 2 diabetes.

DETAILED DESCRIPTION:
The study will last 12-16 weeks and requires 10-13 visits to the General Clinical Research Center on the University Park campus. All food and snacks will be provided for 10 weeks. At the end of each of three diet periods, participants will undergo a test of endothelial function, an oral glucose tolerance test, and a cardiovascular stress reactivity test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, nonsmoking adults, aged 30-75 years (women must be post-menopausal)
* Diagnosed with Type 2 diabetes

Exclusion Criteria:

* Insulin, more than one blood pressure lowering medication, daily aspirin, NSAID therapy, oral steroids within the last 6 weeks, oral contraceptives, and hormone replacement therapy
* Chronic disease such as cardiovascular disease or any complications of diabetes (retinopathy, neuropathy, etc).
* Allergies or aversions to pistachios
* Unwillingness to consume all foods provided and no other meals or snacks for the 10 weeks of diet intervention

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cardiovascular responses to stress | End of each diet period
Insulin sensitivity and resistance | End of each diet period
Lipids and lipoproteins | End of each diet period

SECONDARY OUTCOMES:
Vascular endothelial function | End of each diet period
Mood and perceived stress | End of each diet period

CONTACTS AND LOCATIONS:
Overall Officials: Sheila G. West, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University - General Clinical Research Center, University Park, Pennsylvania, United States

REFERENCES:
- [Background] Gebauer SK, West SG, Kay CD, Alaupovic P, Bagshaw D, Kris-Etherton PM. Effects of pistachios on cardiovascular disease risk factors and potential mechanisms of action: a dose-response study. Am J Clin Nutr. 2008 Sep;88(3):651-9. doi: 10.1093/ajcn/88.3.651. PMID 18779280
- [Derived] Sauder KA, Pokorney PE, McCrea CE, Ulbrecht JS, Kris-Etherton PM, West SG. Noninvasive assessment of hemodynamics: a comparative analysis of fingertip pulse contour analysis and impedance cardiography. Blood Press Monit. 2015 Aug;20(4):209-14. doi: 10.1097/MBP.0000000000000118. PMID 25815738
- [Derived] Sauder KA, McCrea CE, Ulbrecht JS, Kris-Etherton PM, West SG. Pistachio nut consumption modifies systemic hemodynamics, increases heart rate variability, and reduces ambulatory blood pressure in well-controlled type 2 diabetes: a randomized trial. J Am Heart Assoc. 2014 Jun 30;3(4):e000873. doi: 10.1161/JAHA.114.000873. PMID 24980134
- See also: Vascular Health Interventions Lab, Penn State University — http://bbh.hhdev.psu.edu/lab/WestLab/index.html